CLINICAL TRIAL: NCT01243619
Title: 3'-Deoxy-3'(18) F-Fluorothymidine Positron Emission Tomography/Computed Tomography (PET/CT) for Initial Staging, Radiotherapy Target Definition, and Assessment of Response to Therapy in Patients With Esophageal Cancer: A Pilot Study
Brief Title: FLT PET/CT for Staging, Target Definition and Assessment of Response to Therapy in Patients With Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Harvey Mamon, MD, PhD, Radiation Oncologist, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-169
Record Dates: First submitted 2010-09-30; First posted 2010-11-18 (Estimated); Results first posted 2015-03-05 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Esophageal Cancer
Keywords: PET; CT; radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FLT PET (Experimental): This is a single arm trial, in which all patients receive three FDG-PET scans and three FLT-PET scans, before, during and after pre-operative chemoradiation for esophageal cancer.
  Interventions: Drug: 3'-deoxy-3'-(18) F-fluorothymidine

INTERVENTIONS:
Drug: 3'-deoxy-3'-(18) F-fluorothymidine — Radio-tracer for tumor imaging
  Other Names: FLT

SUMMARY:
The purpose of this pilot study is to develop a more advanced software program that will collect, compare and analyze tumor images for evaluation. Another purpose of this study is to learn if a new radio-tracer for tumor imaging called 3'-deoxy-3'(18) F-fluorothymidine (FLT) can improve the evaluation of tumors during a PET/CT scan. This new type of image tracking is meant to improve the visualization of tumor active and size.

DETAILED DESCRIPTION:
* The following are standard medical procedures that are part of regular cancer care that the participant would probably have done even if they did not join the study: Chemotherapy; physical examination; pregnancy test (if applicable); diagnostic FDG-PET/CT scan before and after treatment to evaluate disease.
* The following diagnostic procedures are being done specifically because of this study: Three FLT-PET/CT scans before, during and after treatment and one FDG PET/CT scan during treatment.
* Participants will be in this research study for approximately 12-14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the esophagus or gastroesophageal junction. Biopsy or cytology of the primary tumor, or of involved regional lymph nodes, is acceptable.
* Tumors must be TNM stage T2-4, N0-1, M0 as determined by pretreatment endoscopic ultrasound. T1 tumors are eligible if they are T1, N1, M0. Regional thoracic lymph node involvement is permitted.
* Disease must be clinically limited to the esophagus or gastroesophageal junction. If the tumor extends below the gastroesophageal junction into the proximal stomach, 50% of the tumor must involve the distal esophagus or gastroesophageal junction. Adenocarcinomas of the distal esophagus would therefore include tumors of the gastroesophageal junction which involve equally both the distal esophagus and proximal stomach, or Siewert type II. Tumor much be surgically resectable and have a minimum length of 2cm.
* Patients must be judged by their oncologist to be a candidate for combined modality therapy with chemotherapy consisting of oxaliplatin with protracted infusion 5-FU and concurrent radiation.
* FDG PET/CT performed off-site must be available for review by the Overall PI in DICOM format and has been performed within one month of study entry
* 18 years of age or older
* ECOG Performance Status 0-1
* Laboratory values as outlined in the protocol

Exclusion Criteria:

* No prior chemotherapy or radiotherapy is permitted. Patients must be at least 4 weeks since major surgery, or must have recovered from the effects of minor surgery.
* No prior malignancies (other than basal cell or squamous cell carcinoma of the skin, in situ cervical carcinoma, or superficial transitional cell bladder carcinoma) are permitted unless diagnosed and/or treated 3 years or longer before registration and without evidence of recurrence.
* Patients with the following tumor characteristics are not eligible: TIS (in situ carcinoma); tumors determined to be T1N0 following endoscopic ultrasound; supraclavicular (for distal tumors) or celiac (for proximal tumors) lymph node involvement, as determined by EUS, CT scan, or PET scan, unless this is proven to be a false positive by an appropriate biopsy; cervical esophageal tumors, or gastric cancers with minor involvement of the gastroesophageal junction or distal esophagus; no patients with tracheoesophageal fistulas
* Patients with evidence of metastatic disease
* No poorly controlled diabetes despite attempts to improve glucose control by fasting duration and adjustment of medications
* Pregnant and breast feeding women are excluded
* HIV-positive individuals on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harvey J. Mamon, MD, PhD, Principal Investigator — Dana-Farber/Brigham and Women's Cancer Center
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single arm open label pilot study. Study was expected to enroll five patients at Dana Farber Cancer Institute and Brigham and Women's Hospital. The study was initiated in August 2010 and the primary completion date was March 2013.
Groups:
- All Participants: All participants in the trial received an FDG PET scan before and after chemoradiation for esophageal cancer. In addition, as experimental staging studies, patients on this protocol received a third FDG PET scan during chemoradiation, and received three FLT PET scans before, during and after chemoradiation. All patients received standard of care chemotherapy and radiation and went on to esphagectomy.
Period: Overall Study
Arm/Group | All Participants
Started | 5
Completed | 5 (Patient enrollment is complete, data analysis is ongoing)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Determined by the Number of Participants Who Had All Three Sets of Completed Serial PET Scans That Were Imported for Analysis
Description: Determine the possibility of aquiring three sets of serial Positron emission tomography (PET) scans from 5 patients at designated time points and to develop a mechanism to import and analyze images from F-fluoro-3'-deoxy-3'-L-fluorothymidine (FLT)-PET, Fluorodeoxyglucose(FDG)-PET and Computed Tomography (CT) on a single advanced software platform with deformable image registration capability. We will report patient acceptance of and compliance with this regimen, as well as the utility of the software platform for conducting the proposed analysis.
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- All Participants: All participants in the trial received an FDG PET scan before and after chemoradiation for esophageal cancer. In addition, as experimental staging studies, patients on this protocol received a third FDG PET scan during chemoradiation, and received three FLT PET scans before, during and after chemoradiation. All patients received standard of care chemotherapy and radiation and went on to esphagectomy.
  All patients accepted and complied with having three sets of PET scans performed (six total PET scans).
  The software used in this protocol has allowed quantitative comparison among the PET scans.
Arm/Group | All Participants
Number analyzed (Participants) | 5
participants | 5

2. Other Pre Specified Outcome: Analyze Correlation Between FDG and FLT PET Scans, and the Correlation Between Both Types of PET Scan and the Response to Treatment.
Description: We will compare the findings of FDG and FLT PET scans at pre-treatment, mid-treatment and post-treatment time points to determine how closely they correlate with each other, and if there is a specific time point at which any observed differences between FDG and FLT PET scans are most pronounced. We will also determine which of the six PET scans may correlate most closely with the response to treatment as determined by pathologic findings at esophagectomy.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No